CLINICAL TRIAL: NCT02181179
Title: Examining Yoga's Effects on Aspects Related to Stress and Smoking Behavior
Brief Title: Examining Yoga's Effects on Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014040107
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Yoga; Waitlist
Keywords: yoga; exercise intervention; smoking; stress; mind-body; intervention
MeSH Terms: conditions — Smoking | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga (Active Comparator): This will involve participating in at least two 60-minute Vinyasa yoga sessions each week for eight weeks (weeks 1-8). This will begin the week following a baseline laboratory appointment. These sessions will be conducted at a local Austin studio that has numerous locations in the area.
  Interventions: Behavioral: Yoga
- Waitlist (No Intervention): If randomized to this group, participants will complete weekly assessments only and not yoga during their time in the study. Following full completion of the study (i.e., after week 10), participants will be compensated with a voucher for 2 free months of yoga.

INTERVENTIONS:
Behavioral: Yoga — The yoga intervention will be an 8-week program involving two 60-minute sessions each week at a local studio with three locations in Austin. Participants will be instructed to take classes deemed within a moderate-to-vigorous intensity dose. Participants will also be encouraged both by the PI and yoga instructors to complete the entire 60 minutes of yoga, urged to do only what is comfortable and not push themselves beyond their physical limits.
  Other Names: Hatha yoga; vinyasa yoga
  Arms: Yoga

SUMMARY:
The primary aim of this research study is to examine the effects of an 8-week yoga program on aspects related to nicotine dependence, stress, and coping during a smoking quit attempt.

Guided by initial studies reporting on the effects of yoga on putative mediators of smoking relapse (i.e., cortisol, distress intolerance, withdrawal symptoms), the proposed experiment examines the effects of an 8-week yoga practice on nicotine withdrawal intensity by way of aiding withdrawal characteristics predictive of smoking relapse. The long-term objectives of the proposed line of research are to: (1) inform theoretical models of nicotine withdrawal, (2) guide the development of effective alternative interventions for smokers susceptible to relapse during the critical withdrawal period (i.e., smokers low in distress tolerance), and (3) to help guide behavioral strategies for treating substance addictions broadly.

DETAILED DESCRIPTION:
As the leading cause of preventable death in the US and a major cause for chronic disease/mortality worldwide, smoking represents a major public health issue in need of effective interventions to reduce its burden. The development of such strategies is best directed by basic research on the biobehavioral processes underlying smoking maintenance and relapse. A major predictor of cessation failure is nicotine withdrawal, especially among individuals low in distress tolerance (DT).

Reducing nicotine withdrawal-related distress and relapse in low DT smokers may require the regulation of certain hormones involved in the hypothalamic pituitary axis (HPA-axis) (i.e., the human stress response). Regular practice of yoga, a mindfulness-based form of physical activity, emerges as a promising strategy for regulating the HPA-axis, decreasing withdrawal symptoms, and increasing DT, thus promoting smoking cessation success.

We will randomly assign 50 smokers (≥10 cigarettes daily) low in DT to either an 8-week yoga intervention [YOGA] or a waitlist control [WL] prior to undergoing a self-guided quit attempt. We hypothesize participants assigned to the yoga condition (relative to waitlist) will differ on various outcomes assessed throughout the intervention (e.g., quit status, negative affective states, stress, hormonal changes, withdrawal) and, quit day, and throughout the 2-week quit follow-up period.

More specifically, we hypothesize that certain typical maladaptive, during-withdrawal changes may be attenuated through YOGA. We also hope to obtain initial effect sizes of the advantage of yoga compared to waitlist for point-prevalent abstinence at two weeks following an unaided quit attempt.

ELIGIBILITY:
Inclusion Criteria:

* Female only patients ages 18-65 capable of providing informed consent
* Daily smoker for at least one year.
* Currently smoke an average of at least 10 cigarettes per day.
* Sedentary as defined by moderate-intensity exercise less than 2 days/wk for at least 30 minutes each
* Written physician approval/medical clearance to participate in an exercise/yoga protocol.

-Report motivation to quit smoking of at least 5 on a 10-point Likert-type scale - -Express interest in making a serious, unassisted quit attempt in the next month-

* Have not decreased number of cigarettes smoked in the past 6 months

Exclusion Criteria:

* Use of other tobacco products
* Severe obesity (BMI ≥ 40)
* Currently pregnant or plans to become pregnant
* Diagnosis of a schizophrenia or bipolar-spectrum disorder
* Currently suicidal or suicide high-risk or severe depression
* Use of corticosteroid medications
* Change in medication doses for past 6-months for psychotropic drugs
* Receiving concurrent psychotherapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Measurement of Objective Stress through Hormonal Biomarkers (Hair & Salivary Cortisol) | Collected at pre-and-post intervention (Baseline and Quit day, Week 9)
  we will collect biological samples of hair and saliva to assess changes in biomarkers in response to yoga, and as a potential mechanism by which yoga may aid in smoking cessation. Saliva samples will be collected with Salivettes (Sarstedt, Rommelsdorf, Germany), plastic vials with cotton dental rolls inside. Participants will complete 2 Salivettes at each of three separate 12-hr collection periods. participants will provide two hair strand samples cut by trained personnel (Gerber et al., 2012; Suave et al., 2007; Meyer & Novak, 2012). Hair strands are cut close to the scalp from the posterior vertex of the head using surgical scissors.
Minnesota Nicotine Withdrawal Scale-Revised | post-yoga Week 9 on Quit day and week 10 follow-up
  MNWS-R (Hughes & Hatsukami, 1986) is a validated 15-item self-report measure of withdrawal severity rated on a 5 point Likert scale (0 "none" to 4 "severe") that will establish level of nicotine withdrawal as a major outcome assessed between groups during quit period.

SECONDARY OUTCOMES:
Self reported anxiety sensitivity - Anxiety Sensitivity Scale (ASI). | Weekly from pre-to-post intervention (screen, Baseline, weeks 1-10)
  The 16-item ASI will be employed to assess sensitivity to, and discomfort with, physical anxiety sensations. The ASI (Reiss et al., 1986) as a screening criterion (ASI≥ 20 as indicative of elevated AS) and an outcome measure. The ASI has good internal consistency, test-retest reliability, and excellent convergent validity with other established measures. For the purpose eligibility assessment, this measure will be completed during the Online Prescreen. This measure will also be assessed weekly as a primary outcome assessed between groups.
carbon monoxide (CO) | Screen, week 0 (baseline), week 9 Quit day, & week 10 follow up
  Participants will complete carbon monoxide (CO) analysis of breath sample (≥8ppm cutoff; Jarvis et al., 1987) to determine smoking status during ad-libitum phases and to assess smoking quit status during the quit period.
Smoking point-prevalence - timeline follow back calendar | Weeks Screen, 0 (baseline), 1-8 (intervention), 9-10 (quit period)
  Participants will complete the full timeline follow back calendar (TLFB; past-week) to assess daily point-prevalence of cigarettes both as a screening tool (reflecting ≥ 10 cigarettes/day on average for the past year; and throughout the study period. point prevalence during quit period will be examined between groups and verified with biochemical measurement of lung carbon monoxide (CO)
Five Facet Mindfulness Questionnaire (FFMQ). | Weekly from baseline to post-yoga (week 9)
  The FFMQ (Baer et al., 2006) is a 39-item self-report measure of mindfulness components: observing, describing, acting with awareness, nonjudging of inner experience, and nonreactivity to inner experience. This will be given across intervention to assess changes in response to the mindfulness-based practice of yoga (i.e., with changes compared between groups).
Barratt Impulsiveness Scale (BIS) of Trait Impulsivity | Eligibility Screen
  BIS-15 (Spinella, 2007) is a 15-item self-report measure of 3 non-overlapping impulsivity components: non-planning, motor impulsivity, and attention impulsivity. As one of the most commonly used measures of impulsivity, it has demonstrated validity and reliability in neuropsychiatric and healthy populations. The 15-item short form of the BIS has shown to retain its 3-factor structure when subject to factor analysis and maintained good reliability and validity (Spinella 2007). screening tool (coupled with the ASI) to select individuals scoring above the community norm for impulsivity (Mean score ≥ 32.6 out of 54), as this smoking population may be especially at risk for reactivity to withdrawal symptoms/withdrawal related relapse.
Balloon Analogue Risk Task (BART). | Pre-to-post (at eligibility screen & week 9 visit).
  BART is a laboratory-based behavioral measure of risk taking, evidencing sound experimental properties. It has been shown to predict risk-related constructs (e.g., impulsivity, sensation seeking) as well as self-reported real-world risk behaviors in adults and adolescents (Lejuez et al., 2002). Riskiness on the BART has been correlated with occurrence of addictive, health, and safety risk behaviors, indicating that the BART may be a useful clinical assessment tool. Importantly, as smokers have demonstrated greater total riskiness and sensation seeking on the BART, we will administer the task at pre-and-post intervention as a secondary predictor of smoking outcomes in our trial, possibly indicative of greater difficulty quitting related to impulsivity (which may also be aided with yoga, and thus, differences in behavior will be compared between groups).
Computerized Delay Discounting Task (DDT). | Pre-to-post (eligibility screen & week 9 visit)
  The Delay Discounting choice task is a valid and reliable computer adaptive procedure developed for the purpose of studying choice behavior and delayed reward (Richards et al., 1999). The program asks the participant to decide between a higher amount of money (e.g., $10) to be received after one of the different delay periods (e.g., 1 day, 1 week) or a smaller amount of money (e.g. $1) to be received immediately. Because scores on DDT appear to be related to smoking status and level of nicotine dependence (Sweitzer et al., 2008) this measure was included both as a secondary screening predictor of smoking cessation success, and to observe possible pre-to-post changes afforded by yoga. Changes in behavior on this task will compared between groups.
Distress Tolerance Scale (DTS). | Weekly; Baseline (week 0) through week 10 follow up
  The DTS (Simons & Gaher, 2005), a 15-item self-report measure of physical and psychological distress tolerance, will assess changes in DT; it consists of a 5-point Likert scale with possible ratings ranging from strongly agree to strongly disagree. DTS has high internal consistency (alpha=.82). This will serve as a secondary measurement of distress tolerance, accompanying the ASI, and assessed through between-group changes.
Mood and Anxiety Symptom Questionnaire (MASQ). | Quit day week 9
  The MASQ is a self-report measure derived from the tripartite model (Watson et al., 1995). It includes 62 items rated on a scale ranging from 1 (not at all) to 5 (extremely) focusing on how much an individual has experienced specific affect symptoms in the past week. Four subscales include: Anxious Arousal, Anhedonic Depression, General Distress: Anxious Symptoms, and General Distress: Depressive symptoms. We will use the MASQ to assess affective changes in response to 12-hour withdrawal. The MASQ has been employed in previous smoking cessation work (e.g., Zvolensky et al., 2009), and therefore, beyond being psychometrically sound, offers a higher degree of comparability across research. Ratings will be compared between-groups
Fagerstrom Test of Nicotine Dependence (FTND). | Week 0, 6, 9
  The FTND (Heatherton, Kozlowski, Frecker, & Fagerstrom, 1991) has shown good internal consistency, a single dimension factor structure, and positive relationships with degree of nicotine intake. Dependence status will be assessed at baseline, mid, and post-treatment. This measure will serve to quantify nicotine dependence, which will be used as a covariate in the primary analyses.
Beck Depression Inventory (BDI). | Eligibility screen, weeks 0, 6, 9
  The BDI (Beck, Mendelson, Mock, & Erbaugh, 1961) is a widely used 21-item, self-report inventory designed to measure severity of depressive symptoms. Individuals will only be eligible with scores of ≤30 on the BDI (scores ≥30 indicate severe depression). The BDI will also be administered throughout the protocol to assess changes in depressive symptoms possibly affected through yoga.

CONTACTS AND LOCATIONS:
Overall Officials: Johnna Medina, M.A., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- See also: Anxiety and Health Behaviors Lab — http://labs.la.utexas.edu/smits/study-participation/yogas-effects-on-stress-smoking/